CLINICAL TRIAL: NCT06198452
Title: Vision Improvement for Patients With Age-Related Macular Degeneration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIS #001
Record Dates: First submitted 2023-12-21; First posted 2024-01-10 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vision Improvement (Experimental)
  Interventions: Procedure: Vision Improvement

INTERVENTIONS:
Procedure: Vision Improvement — Laser Vision Improvement for Patients with Age-Related Macular Degeneration

SUMMARY:
This study is being conducted to assess the safety and efficacy of the VIS, LLC (VIS) Opti-K Low Vision Aid Device and treatment to provide vision improvement to patients with age-related macular degeneration.

DETAILED DESCRIPTION:
This study is being conducted to assess the safety and efficacy of the VIS, LLC (VIS) Opti-K Low Vision Aid Device and treatment to provide vision improvement to patients with age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are candidates for this study:

1. Male or Female
2. Any race
3. Patient is at least 50 years old.
4. Patient has diagnosed end stage dry or wet age-related macular degeneration in one or both eyes, as verified by a complete ocular examination.
5. Patient is pseudophakic or is phakic with no clinically significant cataract in eye(s) to be treated.
6. Patient has manifest refraction, spherical equivalent (MRSE) between -1.50 D to 1.50 D in eye(s) to be treated.
7. Patient has moderate to severe vision impairment due to age-related macular degeneration with best spectacle-corrected distance visual acuity (CDVA) of 20/80 or worse (decimal less than or equal to 0.25; logMAR ≥ 0.60).in the better eye.
8. Patient has CDVA of 20/400 or better (decimal greater than or equal to 0.05; logMAR ≤ 1.30) in the worse eye.
9. Patient is not a contact lens (CL) wearer.
10. Patient is willing and able to comply with all examinations.
11. Patient must be competent to sign an informed consent form before study entry.

Exclusion Criteria:

Subjects who meet any of the following criteria are to be excluded from this study:

1. Corneal disease or corneal disorder in either eye.
2. Pathological retinal morphology in either eye that completely affects the entire 10° (3 mm diameter) of the retina centered on the foveola.
3. Gonzalez-Markowitz chart Potential Visual Acuity (PVA) in the eye to be treated that is not improved by at least four lines compared to CDVA;
4. Increased IOP (above 20 mm Hg), glaucoma or history of glaucoma;
5. Previous corneal surgery in the eye to be treated; and
6. Presence or history of any other condition or finding that, in the opinion of the investigator, makes the patient unsuitable as a candidate for study participation or that may confound the outcome of the study.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1 year
  Standard measurements of visual acuity before and after treatment

IPD SHARING:
Plan to Share IPD: No